CLINICAL TRIAL: NCT00909337
Title: Early Therapy of Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-295 ex 06/07
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Pulmonary Hypertension; Systemic Sclerosis
MeSH Terms: conditions — Hypertension, Pulmonary; Scleroderma, Systemic | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosentan (Other): In this study, all participants have normal pulmonary arterial pressure at rest and elevated pulmonary arterial pressure during exercise. First, they were followed up for a year and were controlled after 1 year without specific therapy for pulmonary hypertension. Then Bosentan was introduced. A second control showing the effects of the therapy was done after 6 months. The changes in the "therapy period" can be compared with the changes in the "follow up period".
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — 2x62.5mg for 4 weeks, then 2x125mg
  Other Names: Tracleer

SUMMARY:
Exercise-induced increase of the pulmonary arterial pressure may be an early sign of pulmonary arterial hypertension. It has been shown that patients with normal pulmonary arterial pressure at rest but elevated pulmonary arterial pressure during exercise have a decreased exercise-capacity and may have a worse prognosis compared to patients with normal pulmonary arterial pressure values at rest and during exercise. According to the currently used definition pulmonary hypertension can be diagnosed if the mean pulmonary arterial pressure is higher than 25mmHg at rest or 30mmHg during exercise. In this study patients with a risk for pulmonary arterial hypertension (connective tissue disease) and increased pulmonary arterial pressure values during exercise are receiving a therapy with a dual endothelin receptor antagonist - bosentan, a therapy established for pulmonary arterial hypertension. The therapy effect is than compared to the recorded changes before the introduction of this therapy.

DETAILED DESCRIPTION:
Bosentan is an established therapy in pulmonary arterial hypertension, which may be diagnosed when the mean pulmonary arterial pressure is >25mmHg at rest or >30mmHg at exercise. Bosentan has shown efficacy, if mean pulmonary arterial pressure was elevated at rest. However, there are no data available of the effects of such a therapy, if the mean pulmonary arterial pressure is normal at rest but elevated during exercise. The purpose of this study is to provide additional data on this group of patients. Our hypothesis is that patients with exercise-induced pulmonary hypertension may show a gradual worsening of pulmonary hemodynamics and potentially a development of manifest pulmonary arterial hypertension (elevated resting pulmonary arterial pressure values) without treatment, while the introduction of Bosentan may improve hemodynamics and exercise capacity in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* exercise-induced pulmonary hypertension
* systemic sclerosis

Exclusion Criteria:

* relevant pulmonary obstruction or restriction
* relevant left cardiac disease
* recent changes in medical therapy
* recent major operations
* recent major cardiovascular diseases
* inability to perform exercise

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change of mean pulmonary arterial pressure at 50W under therapy with Bosentan compared to change of mean pulmonary arterial pressure at 50W before the introduction of therapy with Bosentan | 12months before Bosentan therapy vs. at begin of bosentan therapy vs. 6months under bosentan therapy

SECONDARY OUTCOMES:
pulmonary vascular resistance, peak oxygen uptake | 12months before Bosentan therapy vs. at begin of bosentan therapy vs. 6months under bosentan therapy

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Pulmonology, Graz, Austria

REFERENCES:
- [Derived] Kovacs G, Maier R, Aberer E, Brodmann M, Graninger W, Kqiku X, Scheidl S, Troster N, Hesse C, Rubin L, Olschewski H. Pulmonary arterial hypertension therapy may be safe and effective in patients with systemic sclerosis and borderline pulmonary artery pressure. Arthritis Rheum. 2012 Apr;64(4):1257-62. doi: 10.1002/art.33460. Epub 2011 Nov 11. PMID 22127844